CLINICAL TRIAL: NCT02719210
Title: High Volume Plasma Exchange in Children With Acute Liver Failure and Acute on Chronic Liver Failure-A Prospective Pilot Study.
Brief Title: High Volume Plasma Exchange in Children With Acute Liver Failure and Acute on Chronic Liver Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ALF-02
Record Dates: First submitted 2016-02-17; First posted 2016-03-25 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-05

CONDITIONS: Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute | interventions — Sodium Chloride; Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Volume Plasma Exchange with Standard Treatment (Experimental)
  Interventions: Biological: High Volume Plasma Exchange
- Standard Treatment (Active Comparator): Standard Treatment is defined as anti raised Intra-cranial pressure
  1. Elective positive pressure ventilation in hepatic encephalopathy grade 3 or 4 and in those with features of raised ICP (Intra-cranial pressure).
  2. Mannitol
  3. Hypertonic 3% Saline
  Interventions: Drug: Hypertonic 3% saline; Drug: Mannitol; Device: Elective positive pressure ventilation

INTERVENTIONS:
Biological: High Volume Plasma Exchange
  Arms: High Volume Plasma Exchange with Standard Treatment
Drug: Hypertonic 3% saline
  Arms: Standard Treatment
Drug: Mannitol
  Arms: Standard Treatment
Device: Elective positive pressure ventilation
  Arms: Standard Treatment

SUMMARY:
All the children with acute liver failure who are candidates for transplant but have constraints for transplant will be randomized either to receive standard medical therapy or high volume plasma exchange along with standard medical therapy with the aim to assess the effect of high volume plasma exchange on transplant free survival.

ELIGIBILITY:
Inclusion Criteria:

- Children ≥ 10kg with ALF with INR ≥ 4 or INR ≥ 3 with Hepatic Encephalopathy.

Exclusion Criteria:

1. Evidence of active infection (Age specific neutrophilic leucocytosis (ANC) and procalcitonin ≥ 2 and/or focus of active infection
2. Refusal of consent or assent (annexure 3)
3. Liver resections with liver failure
4. Patients with clinical suspicion of irreversible brain injury
5. Patients with acute kidney injury

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Transplant free Survival. | 7 days
Transplant free survival | 30 days

SECONDARY OUTCOMES:
Survival after liver transplant with or without High Volume Plasma Exchange. | 30 days post procedure
Incidence of organ dysfunction (other than liver and Central Nervous System). | 30 days
Number of organs (other than liver and CNS) affected in children with organ dysfunction. | 30 days
Incidence of High Volume Plasma Exchange related complications- Major/Minor. | within 1 month
Change in hemodynamic parameters and Hepatic Encephalopathy (HE) before and after in the High Volume Plasma Exchange group. | 0 day
Change in hemodynamic parameters and Hepatic Encephalopathy (HE) before and after in the High Volume Plasma Exchange group. | 5 days
Change in Laboratory parameters - Bilirubin, INR and Ammonia in control group. | 0 day
Change in Laboratory parameters - Bilirubin, INR and Ammonia- in control group. | 5 day
Change in the levels of IL-6 and TNF alpha (Tumor Necrosis Factor) in HVPE arm from baseline till within 24-hours of the last session of High Volume Plasma Exchange. | within 24-hours of the last session of High Volume Plasma Exchange
Change in the levels of IL-6 and TNF alpha (Tumor Necrosis Factor) in control arm from baseline till 5 days. | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr Arti Pawaria, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided